CLINICAL TRIAL: NCT01546402
Title: Intraoperative Dexamethasone Implant (Ozurdex®) Improves Outcome of Cataract Surgery in Patients With Diabetic Macular Edema
Brief Title: Intraoperative Dexamethasone Implant Improves Outcome of Cataract Surgery With Diabetic Macular Edema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Aniruddha Agarwal, MD, MBBS, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: aniruddha9
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Macular Edema, Cystoid; Vision Disorders; Diabetic Macular Edema; Cystoid Macular Edema Following Cataract Surgery; Cataract
MeSH Terms: conditions — Macular Edema; Vision Disorders; Cataract | interventions — Calcium Dobesilate; Cataract Extraction; Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phacoemulsification with IOL implant (Experimental): This group (Group B) includes patients who will undergo phacoemulsification with intraocular lens implantation. The dexamethasone implant will not be injected at the beginning of cataract surgery. Using a clear corneal incision, continuous curvilinear capsulorhexis, hydrodissection, phacoemulsification and irrigation/aspiration of the cortex will be performed. Foldable intraocular lens will be implanted in the capsular bag. All patients will receive standard postoperative topical steroid (betamethasone 0.1%), antibiotic (moxifloxacin 0.5%) and homatropine (2%) therapy.
  Interventions: Procedure: Cataract surgery
- Phacoemulsification with Ozurdex (Experimental): This group (Group A) includes patients who will undergo phacoemulsification with intraocular lens implantation with intraoperative long acting steroid injection (Ozurdex ®). The dexamethasone implant will be injected at the beginning of cataract surgery, 4mm from the limbus using the specially designed injector. Using a clear corneal incision, continuous curvilinear capsulorhexis, hydrodissection, phacoemulsification and irrigation/aspiration of the cortex will be performed. Foldable intraocular lens will be implanted in the capsular bag. All patients will receive standard postoperative topical steroid (betamethasone 0.1%), antibiotic (moxifloxacin 0.5%) and homatropine (2%) therapy.
  Interventions: Drug: Dexamethasone Drug delivery system (Ozurdex)

INTERVENTIONS:
Drug: Dexamethasone Drug delivery system (Ozurdex) — It is a sustained release intravitreal implant containing 700µg dexamethasone has been approved by the US-FDA (Food and Drug Administration).
  Other Names: Ozurdex
  Arms: Phacoemulsification with Ozurdex
Procedure: Cataract surgery — Using a clear corneal incision, continuous curvilinear capsulorhexis, hydrodissection, phacoemulsification and irrigation/aspiration of the cortex will be performed. Foldable intraocular lens will be implanted in the capsular bag. All patients will receive standard postoperative topical steroid (betamethasone 0.1%), antibiotic (moxifloxacin 0.5%) and homatropine (2%) therapy.
  Other Names: Phacoemulsification
  Arms: Phacoemulsification with IOL implant

SUMMARY:
This study is undertaken to determine the effect of intravitreal long acting dexamethasone implant, (Ozurdex®) in improving outcome of cataract surgery in patients with diabetic macular edema.

Diabetic Macular Edema and cataract constitute important causes of visual impairment in patients with diabetes. Cataract surgery in patients with diabetic retinopathy is associated with progression of retinopathy.

Several modalities such as non-steroidal anti-inflammatory agents, carbonic anhydrase inhibitors, corticosteroids, hyperbaric oxygen, laser photocoagulation and vitrectomy with internal limiting membrane peeling have been tried for managing inflammatory cystoid macular edema.

Intravitreal Triamcinolone Acetonide (TA), a water insoluble steroid, has been shown to reduce the retinal thickness and improve the visual acuity. However, recurrence of macular edema in patients who receive intravitreal TA is a major concern as the patients need multiple repeat injections.

In search for the ideal corticosteroid preparation, a Dexamethasone Posterior Segment Drug Delivery System (Dexamethasone DDS - Ozurdex®, Allergan Inc, Irvine, California) was recently developed. Promising results have been shown in certain patients with persistent diabetic macular edema receiving this intravitreal drug delivery system with improvement in visual acuity

The present study introduces a novel concept of using intraoperative Ozurdex ® implant in patients with diabetes mellitus while undergoing cataract surgery to minimize the worsening of diabetic maculopathy.

DETAILED DESCRIPTION:
Diabetic Macular Edema (DME) and cataract constitute important causes of visual impairment in patients with diabetes mellitus. Cataract surgery in patients with diabetic retinopathy is associated with progression of both retinopathy and maculopathy in nearly 23-57% of cases, thus affecting the final visual outcome. Post-cataract surgery, macular edema may be due to worsening/presence of pre-existing clinically significant macular edema (CSME) or due to development of Irvine Gass Syndrome where cystoid macular edema (CME) occurs in the post operative period and is believed to be inflammatory in origin. Focal/ grid laser photocoagulation is the standard of care in the management of CSME, which may be pre-existing at the time of cataract surgery or worsens following surgery. Several adjuncts including intravitreal corticosteroids, Pegaptanib Sodium (Macugen; Pfizer, New York), Ranibizumab (Lucentis; Genentech, South San Francisco, California), Bevacizumab (Avastin, Genentech) have been tried in an attempt to improve the visual results.

Several modalities such as non-steroidal anti-inflammatory agents, carbonic anhydrase inhibitors, corticosteroids, hyperbaric oxygen, laser photocoagulation and vitrectomy with internal limiting membrane peeling have been tried for managing inflammatory cystoid macular edema13. Intravitreal Triamcinolone Acetonide (TA), a water insoluble steroid, has been shown to reduce the retinal thickness and improve the visual acuity14-16. However, recurrence of macular edema in patients who receive intravitreal TA is a major concern as the patients need multiple repeat injections because of the short half life of the drug (18.6 days). A more potent steroid, dexamethasone has also been tried as an alternative to TA for macular edema; however, its short half life of only 3 hours prevents its clinical application.

In search for the ideal corticosteroid preparation, a Dexamethasone Posterior Segment Drug Delivery System (DDS) - Ozurdex®, Allergan Inc, Irvine, California) was recently developed which has generated new interest in this molecule. It is a sustained release intravitreal implant containing 700µg dexamethasone has been approved by the US-FDA (Food and Drug Administration) for treatment of macular edema in retinal vein occlusions. Promising results have been shown in certain patients with persistent diabetic macular edema receiving this intravitreal drug delivery system with improvement in visual acuity.

The present study introduces a novel concept of using intraoperative Ozurdex ® implant in patients with diabetes mellitus while undergoing cataract surgery to minimize the worsening of diabetic maculopathy.

ELIGIBILITY:
Inclusion Criteria:

The patients of Type 2 Diabetes Mellitus fulfilling the following inclusion criteria shall be enrolled in the study:

1. Presence of visually significant cataract requiring surgery (any grade)
2. Patients with Non-proliferative Diabetic Retinopathy (NPDR) with/without clinically significant macular edema (CSME)
3. Patients with Proliferative Diabetic Retinopathy (PDR) with/without CSME where proliferative component has been adequately treated with laser photocoagulation.

All patients fulfilling criteria 1 with 2 or 3 shall be enrolled in the study. The patients of either sex up to the age of 60 years would be included for the study.

Exclusion Criteria:

The following would be the exclusion criteria:

* Presence of untreated proliferative diabetic retinopathy
* Patients with history of ocular hypertension or glaucoma
* Presence of associated conditions that may exacerbate macular edema, i.e. uveitis, retinal vein occlusions, neovascular glaucoma
* History of use of drugs such as prostaglandin analogues, adrenaline or nicotinic acid
* Patients with post-operative media haze or pupillary non-dilation that does not allow good fundus photography, Fundus Fluorescein Angiography (FFA) and Optical Coherence Tomography (OCT).
* Patients who develop any intraoperative complication including posterior capsular rent, vitreous loss, zonular dehiscence, etc shall be excluded from the study in both the groups

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vishali R Gupta, MBBS MS, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; ANIRUDDHA K AGARWAL, MBBS, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Jagat Ram, MBBS MS, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Amod Gupta, MBBS MS, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phacoemulsification With IOL Implant | Phacoemulsification With Ozurdex
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phacoemulsification With IOL Implant | Phacoemulsification With Ozurdex | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.56 (6.78) | 59.56 (4.64) | 58.56 (5.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in the Central Macular Thickness
Description: The primary outcome is the change in the central macular thickness, either an increase or decrease, as measured by optical coherence tomography as compared to the preoperative thickness.
Time Frame: Baseline and 6 MONTHS
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Phacoemulsification With IOL Implant | Phacoemulsification With Ozurdex
Number analyzed (Participants) | 10 | 10
Microns | 85.67 (101.89) | -18.22 (76.20)

2. Secondary Outcome: Change in the Visual Acuity
Description: Change in the visual acuity as measured by the Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity scale (number of letters at 6 months - number of letters at baseline) The number of letters read on the ETDRS scale will be measured, with 0 being the worst and 35 being the best
Time Frame: Difference in number of letters read (6 months minus baseline)
Measure: Mean (Standard Deviation); unit: Number of letters on ETDRS scale
Arm/Group | Phacoemulsification With IOL Implant | Phacoemulsification With Ozurdex
Number analyzed (Participants) | 10 | 10
Number of letters on ETDRS scale | 0.11 (0.05) | 15.22 (0.023)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Phacoemulsification With IOL Implant | Phacoemulsification With Ozurdex
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No